CLINICAL TRIAL: NCT04151979
Title: MRI for the Diagnosis of Placenta Accreta Spectrum
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: PAS001
Record Dates: First submitted 2019-10-24; First posted 2019-11-05 (Actual); Last update posted 2019-11-05 (Actual); Status verified 2019-10

CONDITIONS: Placenta Accreta
Keywords: placenta accreta spectrum; MRI; score scale; diagnosis
MeSH Terms: conditions — Placenta Accreta; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Placenta Accreta Spectrum (PAS) is a disease associated with abnormal placental adhesion and invasion. In recent years, the incidence of PAS has increased significantly, which can cause massive postpartum hemorrhage, hysterectomy,and even maternal mortality. The research team of Peking university third hospital developed the ultrasound rating scale in china at first to conduct preliminary assessment of the PAS risk which can identify the severity of cases. In a basis of ultrasound, plan to explore the MRI for the the investigators diagnosis of PAS according to some specific PAS features, like the the uneven signal intensity , the myometrial discontinuity, and black band on T2 image, and finally established a MRI scoring system of PAS. MRI score system of PAS can reduce the subjective difference of the clinician's visual reading, and assist the clinician to assess the risk of sever PAS further, and conduct perioperative preparation to reduce the risk of maternal morbidity and mortality to achieve a better clinical outcome.

DETAILED DESCRIPTION:
Placenta Accreta Spectrum (PAS) is a disease associated with abnormal placental adhesion and invasion. In recent years, the incidence of PAS has increased significantly, and the main risk is high hysterectomy rate,massive postpartum hemorrhage, and even maternal mortality in women at childbearing age. The research team of Peking university third hospital developed the ultrasound rating scale in china at first to conduct preliminary assessment of the PAS risk which can identify the severity of cases and guide the junior hospitals to transfer. Peking University third hospital is in the leading position in the preoperative diagnosis of PAS currently.

Magnetic resonance imaging (MRI) has become a common method for preoperative evaluation for sever cases. MRI can provide a map of the placenta and PAS features, like the uterus enlarged significantly, the uneven signal intensity , the myometrial discontinuity, and black band on T2 image. It has a high diagnostic value. At present, only Lim and Ueno reported MRI scoring system for PAS. Due to the small sample size and the limitation of the research methods, a widely applicable rating scale has not been established. MRI score system of PAS can reduce the subjective difference of the clinician's visual reading, and assist the clinician to assess the risk of sever PAS further, and conduct perioperative preparation to reduce the risk of maternal morbidity and mortality and achieve a better clinical outcome.

ELIGIBILITY:
Inclusion Criteria:

1. Patients diagnosed as scarred uterus(with a history of cesarean section)
2. "ultrasound score" of PAS≥ 6 points who undergo MRI
3. Terminate pregnancy or childbirth in Peking university third hospital. -

Exclusion Criteria:

1. Patients who didn't undergo MRI
2. Patients who didn't deliver the baby in PUTH -

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The patients who have risk factors of PAS, undergo "ultrasound scoring" and MRI ,finally delivered in Peking university third hospital.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2015-01-01 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Rate of PAS diagnosed | one week after surgery
  diagnose as PAS through clinical observation or specimen pathology after surgery

SECONDARY OUTCOMES:
Blood loss volume(ml) | 24 hours after surgery
  The blood loss volume during the 24 hours after surgery
Rate of hysterectomy | two weeks after surgery
  Number of patients who were performed hysterectomy/Number of patients with PAS
Rate of preterm labor | two weeks after surgery
  The number of patients who delivered between 28 to 36+6 weeks/Number of patients with PAS
Blood transfusion volume(ml) | two weeks after surgery
  the volume of blood transfusion

CONTACTS AND LOCATIONS:
Overall Officials: YangYu Zhao, MD, Study Director — Peking University Third Hospital
Locations (1):
- Peking University Third Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No